CLINICAL TRIAL: NCT05889416
Title: The Effect of Audit and Feedback Within a National Registry and Implementation Support on Guideline Adherence and Patient Outcomes in Cardiac Rehabilitation: an Open-label Cluster-randomized Effectiveness-implementation Hybrid Trial
Brief Title: The Perfect-CR Implementation Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Margret Leosdottir, Senior Cardiology Consultant, Associate Professor, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Perfect-CR V2.0 2023
Record Dates: First submitted 2023-03-23; First posted 2023-06-05 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Infarction; Risk Reduction
Keywords: Myocardial infarction; Cardiac rehabilitation; Secondary prevention; Audit; Implementation; Practice facilitation
MeSH Terms: conditions — Myocardial Infarction; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Open-label Cluster-randomized Effectiveness-implementation Hybrid Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Implementation of national guidelines on secondary prevention according to local plan and preferences
- Audit and feedback (Active Comparator): Audit and feedback on implementation of national guidelines on secondary prevention through the national quality registry SWEDEHEART
  Interventions: Other: Audit and feedback through a quality registry
- Implementation support (Active Comparator): Audit and feedback through the national quality registry SWEDEHEART and structured implementation support for implementation of national guidelines on secondary prevention
  Interventions: Other: Audit and feedback through a quality registry; Other: Implementation support

INTERVENTIONS:
Other: Audit and feedback through a quality registry — Centres answer CR process and structure variables through the SWEDEHEART registry every six months for three years. Feedback will be accessible online and through annual reports, enabling comparisons with own prior and other centres´ results.
  Arms: Audit and feedback; Implementation support
Other: Implementation support — On-site support to implement guidelines on secondary prevention applying practice facilitation - a multifaceted approach carried out by CR experts who enable personnel at intervention centres to address and overcome challenges in implementing guidelines.
  Arms: Implementation support

SUMMARY:
The goal of this open-label cluster-randomized effectiveness-implementation hybrid trial is to study whether a) audit and feedback of cardiac rehabilitation service delivery within a national quality registry and b) structured implementation support can improve center-level adherence to guidelines and short and long-term patient-level outcomes.

DETAILED DESCRIPTION:
Administering secondary prevention via structured cardiac rehabilitation (CR) programs for patients who have suffered a myocardial infarction (MI) reduces mortality and morbidity and improves quality of life. Still, treatment goal achievement at patient-level and service delivery at center-level are sub-optimal and there is a large variation in program structure and delivery at center-level.

Using an open-label cluster-randomized effectiveness-implementation hybrid trial design, the primary objective of this study is to prospectively evaluate whether a) audit and feedback of CR processes and structures within the national cardiac registry SWEDEHEART and b) supporting CR centers in implementing CR guidelines can increase center-level guideline adherence. The secondary objectives are the following:

* At baseline, to cross-sectionally evaluate the association between center-level adherence to guidelines and patient-level outcomes
* To prospectively study whether audit and feedback of CR processes and structures within the SWEDEHEART registry can improve short- and long-term patient-level outcomes
* To prospectively evaluate whether supporting CR centers in implementing CR guidelines can improve short- and long-term patient-level outcomes
* To evaluate the acceptability, adoption, fidelity, implementation cost, and cost effectiveness of the implementation support

All CR centers in Sweden (approximately 75 centers) will be offered participation in the study. Collectively these centers attend to approximately 8000 patients/year. Patient-level outcome data will be retrieved from national registries.

ELIGIBILITY:
Centre-level

Inclusion Criteria:

* Centres report to the SWEDEHEART registry

Exclusion Criteria:

* Unwillingness to participate in the study

Patient-level

Inclusion Criteria:

* Diagnosis of a type 1 MI registered in the SWEDEHEART registry
* Age 18-79 years at discharge from hospital
* Attended at least two follow-up visits at CR centres included in the study

Exclusion Criteria:

* None

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Adherence score | 3 years
  The adherence score reflects center-level adherence to CR processes and structures as recommended in national guidelines on secondary prevention. The score is derived from 39 variables capturing guideline-directed CR structure and processes collected on center-level through the national cardiac registry SWEDEHEART. The score ranges from 0 (worst) to 39 (best).

SECONDARY OUTCOMES:
Blood pressure target attainment | One year
  For patients <70 years of age <130/80 mmHg and for patients ≥70 years <140/80 mmHg (yes/no)
Systolic blood pressure | One year
  Continuous variable in mmHg
Low-density lipoprotein cholesterol target attainment | One year
  <1.4 mmol/L (yes/no)
Low-density lipoprotein cholesterol | One year
  Continuous variable in mmol/L
Self-reported quality of life | One year
  Measured using EuroQoL-Visual Analogue Scale (EQ-VAS) - a vertical visual analogue scale with a range of values between 100 (best imaginable health) and 0 (worst imaginable health)
Self-reported smoking status | One year
  Never smoker, former smoker (>1 month) or current smoker
Self-reported dietary habits | One year
  Dietary habits are assessed by self-report through four questions covering intake of fruit, vegetables, fish and sweets. Each question gives points ranging from 0 (worst) to 3 (best), summing up to a total score of 0-12 points.
Self-reported physical activity | One year
  Number of days during the last week the patient has been physically active for a minimum of 30 minutes (at least 10 minutes at a time) with activity causing shortness of breath and a slightly increased pulse, corresponding to a brisk walk. Permissible values can thus range from 0 days (worst) to 7 days (best).
Attendance in an exercise-based CR programme | One year
  Attended for at least 3 months (yes/no)
Major adverse cardiovascular events (MACE) | Five years
  A composite endpoint of the following events:
  * cardiovascular mortality
  * non-fatal MI
  * non-fatal ischemic stroke
  * coronary revascularization
  * hospitalization for new or worsening heart failure
Total mortality | Five years
  Death from any cause.
Acceptability of the implementation support | Assessed at the time of implementation
  Acceptability reflects the degree to which the intervention is perceived as being feasible, desirable, and appropriate by stakeholders (healthcare providers, i.e., the CR team and organizational leaders) and the level of preparedness of the organization to adopt the intervention. Acceptability will be assessed through semi-structured interviews with healthcare personnel at centers subject to the implementation intervention. Interview guides, allowing for flexibility in terms of order and form of questions and topics, using mainly open-ended and neutral questions will be developed. The exact number of interviews will be decided on after start of the study and will continue until a) no new concepts or categories are identified and b) when there is no need for further elaboration of these.
Adoption of the implementation support | Assessed six months after the implementation support has been provided
  Adoption determines the extent to which the intervention is used in practice. Adoption of the implementation support will be assessed through semi-structured interviews with healthcare personnel at centers subject to the implementation intervention.
Fidelity of the implementation support | Assessed six months after the implementation support has been provided
  Fidelity reflects the degree to which the implementation used in practice adheres to the original design of the intervention. Fidelity will be assessed through semi-structured interviews with healthcare personnel at centers subject to the implementation intervention.
Implementation cost and cost effectiveness | Assessed at the time of implementation
  Reflects resources required to implement the intervention, including the cost of material, staff, and any other expenses incurred as a result of the implementation of the intervention. Based on the cost estimates and the effect of the implementation assistance on patient outcomes, the economic evaluation will then be able to calculate cost-effectiveness ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Margret Leosdottir, Principal Investigator — Skane University Hospital Malmö
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
The data to be used in this study is based on the SWEDEHEART registry. Access to data from the registry needs to be applied for and third-party data usage is not allowed, irrespective of whether the data contain potentially identifying or sensitive data or not. Instead, given ethical study approval from the Swedish Ethical Review Authority, access to SWEDEHEART data can be applied for from the Uppsala Clinical Research Center (UCR) in Sweden. Further information can be found on the UCR www.ucr.uu.se/en/ and Swedish Ethical Review Authority etikprovningsmyndigheten.se/ websites.

REFERENCES:
- [Derived] Michelsen HO, Lidin M, Back M, Duncan TS, Ekman B, Hagstrom E, Hagglund M, Lindahl B, Schlyter M, Leosdottir M. The effect of audit and feedback and implementation support on guideline adherence and patient outcomes in cardiac rehabilitation: a study protocol for an open-label cluster-randomized effectiveness-implementation hybrid trial. Implement Sci. 2024 May 24;19(1):35. doi: 10.1186/s13012-024-01366-8. PMID 38790045